CLINICAL TRIAL: NCT00078351
Title: The Effects of Viscosupplementation Using Synvisc in Symptomatic Osteoarthritis of the Temporomandibular Joint
Brief Title: Synvisc to Treat Osteoarthritis of the Temporomandibular Joint
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040111; 04-D-0111
Record Dates: First submitted 2004-02-23; First posted 2004-02-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Osteoarthritis
Keywords: Chronic Pain; Synvisc; Temporomandibular Joint; Osteoarthritis; TMD; Temporomandibular Joint Osteoarthritis; TMJ OA; Temporomandibular Joint Disease; TMJ
MeSH Terms: conditions — Osteoarthritis; Chronic Pain; Temporomandibular Joint Disorders | interventions — hylan; Injections

INTERVENTIONS:
Procedure: High molecular weight hylan (Synvisc) injection

SUMMARY:
This study will examine the effectiveness of injected hylan (Synvisc) for treating pain associated with osteoarthritis of the temporomandibular joint (jaw joint) and improving function of the joint. Hylan is a synthetic product very similar to a component of normal healthy joint fluid (synovial fluid), which is present in much lower quantities and is abnormal in osteoarthritis. Hylan injections have been beneficial in treating osteoarthritis of the knee.

Patients with temporomandibular (TMJ) joint pain of at least 3 months duration who have mouth opening limitation and moderate to severe joint pain made worse by joint movement may be eligible for this study. Patients must not have any TMJ growth disturbances and must not have had any TMJ surgery for 6 months before entering the study. Candidates are screened with questionnaires, a medical history, and a physical examination of the TMJs, including x-rays and magnetic resonance imaging.

Participants are randomly assigned to receive three injections, each a week apart, of either Synvisc or placebo (a salt-water solution) into the affected joint. Before the first injection, a sample of synovial fluid is collected from the joint by needle aspiration for laboratory analysis. Patients return for follow-up visits 3, 6, and 12 months after the last treatment for a clinical examination of the jaw joint and review of jaw joint symptoms. A second aspiration is requested at the 3-month visit, but is not mandatory. All injections and aspirations are done after anesthetizing the overlying skin and joint capsule to minimize pain or discomfort. Participants record their daily use of pain relief medication throughout the study.

DETAILED DESCRIPTION:
The proposed clinical trial will evaluate the effects of high molecular weight hylan (Synvisc) injection in comparison with control treatment (saline injection) for osteoarthritis (OA) affecting the temporomandibular joint (TMJ). Patients with TMJ OA of at least three-month duration and who have not responded to conservative treatments will be included. Patients will be randomly assigned to either high molecular hylan injection or control. At baseline and follow up visits, clinical outcome measures will be assessed such as pain and range of motion. Positive findings in clinical outcome measures will provide evidence for the clinical utility of Synvisc in patients with painful TMJ OA. In addition to clinical outcome measures, a sample of synovial fluid from the affected joint will be obtained at the baseline visit and at 12 week follow up, and levels of tumor necrosis factor alpha (TNF alpha), Matrix metalloproteinase (MMP) and Tissue inhibitor of metalloproteinase (TIMP) will be analyzed. By studying the synovial fluid levels of TNF alpha, MMP and TIMP, we will assess the effects of viscosupplementation with Synvisc on the local inflammatory process and proteolytic activity in TMJ OA in comparison with control treatment. Positive findings in clinical symptoms and synovial fluid analysis will also provide implications of clinical utility of Synvisc in patients with painful TMJ OA. Furthermore, this analysis of synovial fluid may identify biomarkers associated with OA affecting the TMJ.

ELIGIBILITY:
INCLUSION AND EXCLUSION CRITERIA:

We will recruit patients with TMJ OA defined by the Research Diagnostic Criteria. Patients are required to have chronic preauricular pain for more than 3 months, even though they have received some palliative treatment (NSAIDs and/or stabilization splint therapy). Radiological imaging is indicated in addition to clinical evaluation to confirm the diagnosis of TMJ OA. Radiographic evidence of OA includes flattening of condyle, increased opacity of cortical bone of condyle, or osteophyte formation. Prior to being admitted to the study, patients will be screened with standard temporomandibular joint radiological imaging, including panoramic, tomographic and magnetic resonance imaging (MRI) studies. Radiological imaging will not be repeated at the end of the study unless medically indicated. The patients are required to have mouth opening limitation (less than normal) and moderate to severe joint pain aggravated by jaw movement. Patients who have undergone any TMJ surgery within the preceding 6 months will be excluded, as well as those who have taken analgesic, anti-inflammatory, steroids or narcotic medications during the last 15 days. Further exclusion criteria will be patients who have any TMJ growth disturbances. Patients with red, hot, swollen, tender TMJ, or those with history consist of infectious arthritis, crystal induced arthropathies, and musculoskeletal disorders will also be excluded. Patients with rheumatic disease will also be excluded, this will be determined by baseline blood tests (CBC, chem. 7, ESR, Rheumatoid factor).

Patients will be screened for any positive history of liver or kidney dysfunctions. Any patients with a medical history of diabetes, congestive heart failure, any chronic infections will also be excluded. Subjects that have primary psychiatric disease or score above average in comparison with normative scores on Symptom Checklist (SCL-90R) will not be able to participate. Pregnant women will not be included in the study, this will be determined by a pregnancy test, and subjects will be required to use 2 forms of contraception for the first 3 weeks of the study (to cover the synvisc injections). It is a standard practice in chronic pain study not to include patients who are involved in litigation. Patients with sepsis or with known hypersensitivity to hyaluronan and any of its components will be excluded to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-02; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Huskisson EC, Donnelly S. Hyaluronic acid in the treatment of osteoarthritis of the knee. Rheumatology (Oxford). 1999 Jul;38(7):602-7. doi: 10.1093/rheumatology/38.7.602. PMID 10461471
- [Background] Gabriel SE, Jaakkimainen L, Bombardier C. Risk for serious gastrointestinal complications related to use of nonsteroidal anti-inflammatory drugs. A meta-analysis. Ann Intern Med. 1991 Nov 15;115(10):787-96. doi: 10.7326/0003-4819-115-10-787. PMID 1834002
- [Background] Allison MC, Howatson AG, Torrance CJ, Lee FD, Russell RI. Gastrointestinal damage associated with the use of nonsteroidal antiinflammatory drugs. N Engl J Med. 1992 Sep 10;327(11):749-54. doi: 10.1056/NEJM199209103271101. PMID 1501650